CLINICAL TRIAL: NCT04398095
Title: Hyperthermia and Radiotherapy in the Treatment for In-field Recurrent and Radiation-induced Soft Tissue and Bone Sarcomas
Brief Title: Radiotherapy With Hyperthermia in Recurrent and Radiation-Induced Sarcomas
Acronym: HOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOT1
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2020-05

CONDITIONS: Radiation Induced Neoplasms; Radiation-Induced Cancer; Recurrent Sarcoma; Recurrent Soft Tissue Sarcoma
MeSH Terms: conditions — Neoplasms, Radiation-Induced; Sarcoma | interventions — Radiation Dose Hypofractionation; Diathermy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Radiotherapy with hyperthermia in resectable sarcomas (Experimental): 12x 3 Gy (4 fractions per week) + hyperthermia (6x) + surgery
  Interventions: Radiation: Hypofractionated radiotherapy; Other: Hyperthermia
- Radiotherapy with hyperthermia in non-resectable sarcomas (Experimental): 12x 3 Gy with simultaneous integrated boost 3.5 Gy (4 fractions per week) + hyperthermia (6x)
  Interventions: Other: Hyperthermia; Radiation: Hypofractionated radiotherapy with boost

INTERVENTIONS:
Radiation: Hypofractionated radiotherapy — Resectable or marginally resectable tumors: preoperative hypofractionated 12x 3 Gy radiotherapy (4 days in a week, three weeks) prescribed on planned target volume (tumor volume + elective margins + setup/error margin) with daily image guidance with cone beam-CT or kV-portal position verification.
  Arms: Radiotherapy with hyperthermia in resectable sarcomas
Other: Hyperthermia — Deep hyperthermia (Celsius TCS or BSD-2000) according to local protocol combined with radiotherapy, twice a week.
Radiation: Hypofractionated radiotherapy with boost — Non-resectable/inoperable tumors: definitive hypofractionated 12x 3 Gy radiotherapy prescribed on planned target volume (tumor volume + elective margins + setup/error margin) with simultaneous integrated boost 3.5 Gy per fraction prescribed on boost planned target volume (tumor volume + setup/error margin), 4 days in a week, three weeks.
  Radiotherapy with daily image guidance with cone beam-CT or kV-portal position verification.
  Arms: Radiotherapy with hyperthermia in non-resectable sarcomas

SUMMARY:
After a screening, which consists of biopsy, physical examination, initial diffusion-weighted magnetic resonance imaging (DWI-MRI) or body computed tomography (CT) scan, blood tests and case analysis on Multidisciplinary Team (MDT) meeting, a patient with radiation-induced or in-field recurrent sarcoma will receive the hypofractionated radiotherapy with deep hyperthermia (twice a week) within three weeks. The response analysis in CT or DWI-MRI and toxicity assessment will be performed after 6 weeks. In resectable tumors, a patient will be referred to surgery. In the case of unresectability, the patient will followed-up.

DETAILED DESCRIPTION:
Due to the rarity of radiation-induced (RIS) or previously irradiated recurrent (PIRS) sarcomas, no guidelines nor randomized prospective clinical trials on this topic exist. Thus the management of RIS and PIR is challenging. The only curable modality in non-metastatic RIS/PIRS is radical resection with wide negative margins. The role of secondary radiotherapy in locally advanced RIS/PIRS is unclear, mostly due to the concerns about possible severe side effects after re-irradiation.

The addition of deep hyperthermia to irradiation and in the prolonged gap between the end of moderately hypofractionated radiotherapy (with or without integrated boost) and surgery may allow obtaining the long-term local control with the maintenance of a good treatment tolerance Hyperthermia is a method of increasing the temperature in the tumor to damage cancer cells with minimum injury to the normal cells. It should be combined with another treatment modality (radio- or chemotherapy) rather than used alone. Its efficacy was proven in clinical trials. Treatment tolerance is usually very good.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Eastern Cooperative Oncology Group performance status 0 - 2
* Age ≥18 years old
* Histologically-proven diagnosis of radiation-induced or recurrent soft tissue sarcoma
* Previous radiotherapy within the planned target volume

Exclusion Criteria:

* Histologic diagnosis of rhabdomyosarcoma (except spindle cell and pleomorphic subtype), osteogenic sarcoma, Ewing's sarcoma/PNET, aggressive fibromatosis
* Contraindications to radiotherapy or hyperthermia
* Predicted unacceptable high risk of reirradiation-related toxicity, in the Investigator's judgment
* Unresectable metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Ratio of late adverse events | 18 months
  Ratio of grade 3 or higher late adverse events related to reirradiation, according to CTCAE 5.0

SECONDARY OUTCOMES:
Local control rate | 18 months
Progression-free survival | 18 months
Cancer-specific survival | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Mateusz J Spałek, MD PhD, Principal Investigator — The Maria Sklodowska-Curie National Research Institute of Oncology in Warsaw
Locations (1):
- The Maria Sklodowska-Curie National Research Institute of Oncology in Warsaw, Warsaw, Mazovian, Poland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR

REFERENCES:
- [Background] de Jong MA, Oldenborg S, Bing Oei S, Griesdoorn V, Kolff MW, Koning CC, van Tienhoven G. Reirradiation and hyperthermia for radiation-associated sarcoma. Cancer. 2012 Jan 1;118(1):180-7. doi: 10.1002/cncr.26252. Epub 2011 Jun 28. PMID 21713762
- [Background] Haas RL, Miah AB, LePechoux C, DeLaney TF, Baldini EH, Alektiar K, O'Sullivan B. Preoperative radiotherapy for extremity soft tissue sarcoma; past, present and future perspectives on dose fractionation regimens and combined modality strategies. Radiother Oncol. 2016 Apr;119(1):14-21. doi: 10.1016/j.radonc.2015.12.002. Epub 2015 Dec 21. PMID 26718153
- [Background] Kosela-Paterczyk H, Szacht M, Morysinski T, Lugowska I, Dziewirski W, Falkowski S, Zdzienicki M, Pienkowski A, Szamotulska K, Switaj T, Rutkowski P. Preoperative hypofractionated radiotherapy in the treatment of localized soft tissue sarcomas. Eur J Surg Oncol. 2014 Dec;40(12):1641-7. doi: 10.1016/j.ejso.2014.05.016. Epub 2014 Sep 20. PMID 25282099
- [Background] Lindner LH, Issels RD. Hyperthermia in soft tissue sarcoma. Curr Treat Options Oncol. 2011 Mar;12(1):12-20. doi: 10.1007/s11864-011-0144-6. PMID 21360087
- [Background] Borghede G, Hedelin H. Radiotherapy of localised prostate cancer. Analysis of late treatment complications. A prospective study. Radiother Oncol. 1997 May;43(2):139-46. doi: 10.1016/s0167-8140(96)01871-3. PMID 9192958